CLINICAL TRIAL: NCT05593445
Title: A Phase 2, Randomized, Double-Blind, Vehicle-Controlled, Study of the Efficacy and Safety of Ruxolitinib Cream in Participants With Lichen Sclerosus
Brief Title: A Study to Evaluate the Efficacy and Safety of Ruxolitinib Cream in Participants With Lichen Sclerosus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INCB 18424-220
Expanded Access: NCT03147742 (Approved for marketing)
Record Dates: First submitted 2022-10-21; First posted 2022-10-25 (Actual); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-08

CONDITIONS: Lichen Sclerosus
Keywords: Lichen Sclerosus; Skin Diseases; 18424; Ruxolitinib; topical cream; vulvar disease
MeSH Terms: conditions — Lichen Sclerosus et Atrophicus; Skin Diseases; Vulvar Diseases

STUDY DESIGN:
Intervention Model Description: Study will be a 12 week double-blind period followed by a 12 week open label period.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ruxolitinib cream (Experimental): Ruxolitinib 1.5% cream BID for 12 weeks followed by ruxolitinb 1.5% cream BID (or QD) for 12-weeks in an open-label extension.
  Interventions: Drug: Ruxolitinib cream; Drug: Vehicle cream
- Vehicle Cream (Placebo Comparator): Vehicle cream BID for 12 weeks followed by ruxolitinb 1.5% cream BID (or QD) for 12-weeks in an open-label extension.
  Interventions: Drug: Vehicle cream

INTERVENTIONS:
Drug: Ruxolitinib cream — Ruxolitinib cream is a topical formulation applied as a thin film to affected areas.
  Other Names: INCB018424 cream
  Arms: Ruxolitinib cream
Drug: Vehicle cream — Vehicle cream is matching in appearance to ruxolitinib cream and is to be applied in the same manner as ruxolitinib cream.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Ruxolitinib cream in participants With Lichen Sclerosus. This is randomized, double-blind, vehicle-controlled (DBVC) study with a DBVC period of 12 weeks followed by an open label period (OLE) period of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven LS in the anogenital area.
* Baseline IGA score ≥ 2 for LS.
* Baseline Itch NRS score ≥ 4 in anogenital area.
* Willingness to avoid pregnancy.

Exclusion Criteria:

* Participants who do not have LS involving anogenital area.
* Concurrent conditions and history of other diseases:

  1. Are suspected clinically (or confirmed diagnostically) of having alternative causes of vaginal symptoms including: candidiasis, chlamydia trachomatis, trichomonas vaginalis, neisseria gonorrhoeae, bacterial vaginosis, or herpes simplex.
  2. Have active genital/vulvar lesions at screening and Day 1, not related to LS
  3. Chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 2 weeks before baseline.
* Laboratory values outside of the protocol-defined criteria
* Pregnant or lactating participants or those considering pregnancy during the period of their study participation..
* Other exclusion criteria may apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females aged 18 years or older at screening with a biopsy confirmed diagnosis of Lichen Sclerosus
Enrollment: 61 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haq Nawaz, MD, Study Director — Incyte Corporation
Locations (14):
- United States (12):
  - Cahaba Dermatology, Birmingham, Alabama
  - Mayo Clinic - Scottsdale, Scottsdale, Arizona
  - UC Irvine, Irvine, California
  - The Centers For Vulvovaginal Disorders, Washington D.C., District of Columbia
  - New Age Medical Research Corporation, Miami, Florida
  - Circuit Clinical, West Seneca, New York
  - Unc Dermatology and Skin Cancer Center At Southern Village, Chapel Hill, North Carolina
  - Apex Dermatology, Ashtabula, Ohio
  - Bexley Dermatology, Bexley, Ohio
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Utah Health Care Midvalley Health Center Dermatology, Murray, Utah
  - Seattle Skin and Laser Clinic, Seattle, Washington
- Canada (2):
  - K. Papp Clinical Research, Waterloo, Ontario
  - Clinique Rsf, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 61 participants were randomized into the study. All randomized participants (Intent-to-Treat Population) applied study drug at least once (Safety Population), and 56 participants applied ruxolitinib 1.5% cream at least once during the Open-label Extension (OLE) Period (OLE-Evaluable Population).
Groups:
- Double-Blind, Vehicle-Controlled (DBVC) Period: Ruxolitinib Cream 1.5% BID: Participants applied ruxolitinib 1.5% cream twice daily (BID) for 12 weeks.
- DBVC Period: Vehicle Cream BID: Participants applied matching vehicle cream BID for 12 weeks.
- Open-Label Extension Period: Ruxolitinib Cream 1.5% BID: Participants who completed the Week 12 assessments with no safety concerns could continue into the 12-week Open-label Extension Period. Participants who applied ruxolitinib cream 1.5% BID during the Double-blind, Vehicle-controlled Period continued to apply ruxolitinib cream 1.5% BID for an additional 12 weeks in the Open-label Extension Period. Participants could have cycled between once daily (QD) or BID application of ruxolitinib 1.5% cream based on the investigator's clinical judgment of disease activity.
- Open-Label Extension Period: Vehicle Cream to Ruxolitinib Cream 1.5% BID: Participants who completed the Week 12 assessments with no safety concerns could continue into the 12-week Open-label Extension Period. Participants who applied vehicle cream BID during the Double-blind, Vehicle-controlled Period applied ruxolitinib cream 1.5% BID for 12 weeks in the Open-label Extension Period. Participants could have cycled between QD or BID application of ruxolitinib 1.5% cream based on the investigator's clinical judgment of disease activity.
Period: 12-Week DBVC Period
Arm/Group | Double-Blind, Vehicle-Controlled (DBVC) Period: Ruxolitinib Cream 1.5% BID | DBVC Period: Vehicle Cream BID | Open-Label Extension Period: Ruxolitinib Cream 1.5% BID | Open-Label Extension Period: Vehicle Cream to Ruxolitinib Cream 1.5% BID
Started | 31 | 30 | 0 | 0
Completed | 29 | 27 | 0 | 0
Not Completed | 2 | 3 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Did Not Meet Eligibility Criteria | 1 | 0 | 0 | 0
Period: 12-Week Open-Label Extension Period
Arm/Group | Double-Blind, Vehicle-Controlled (DBVC) Period: Ruxolitinib Cream 1.5% BID | DBVC Period: Vehicle Cream BID | Open-Label Extension Period: Ruxolitinib Cream 1.5% BID | Open-Label Extension Period: Vehicle Cream to Ruxolitinib Cream 1.5% BID
Started | 0 | 0 | 29 | 27
Completed | 0 | 0 | 26 | 25
Not Completed | 0 | 0 | 3 | 2
Not completed — Adverse Event | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- DBVC Period: Ruxolitinib Cream 1.5% BID: Participants applied ruxolitinib 1.5% cream twice daily (BID) for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | DBVC Period: Ruxolitinib Cream 1.5% BID | DBVC Period: Vehicle Cream BID | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (11.28) | 61.9 (12.25) | 60.9 (11.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 30 | 61
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 28 | 25 | 53
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 5 | 5
  White | 31 | 25 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With ITCH4 at Week 12
Description: ITCH4 response was defined as a ≥4-point improvement from Baseline in by-visit Itch Numeric Rating Scale (NRS) score. The Itch NRS is a daily participant-reported measure (24-hour recall) of the worst level of itch intensity. Participants rated itch severity of their lichen sclerosus by selecting a number from 0 (no itch) to 10 (worst imaginable itch) that best described the worst level of itch they experienced in the past 24 hours.
Time Frame: Baseline; Week 12
Population: Intent-to-Treat (ITT) Population: all randomized participants. Treatment groups were defined according to the treatment assignment at the time of randomization regardless of the actual study drug the participant might have taken. Only those participants with a Baseline ITCH NRS Score ≥4 were analyzed. Missing post-baseline values were imputed as Non-Responders at Week 12.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | DBVC Period: Ruxolitinib Cream 1.5% BID | DBVC Period: Vehicle Cream BID
Number analyzed (Participants) | 28 | 30
percentage of participants | 35.7 [18.6 to 55.9] | 40.0 [22.7 to 59.4]
Statistical Analysis 1: Comparison: DBVC Period: Ruxolitinib Cream 1.5% BID vs DBVC Period: Vehicle Cream BID; Test type: Superiority; p = 0.737, Chi-squared; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.29 to 2.41]
Statistical Analysis 2: Comparison: DBVC Period: Ruxolitinib Cream 1.5% BID vs DBVC Period: Vehicle Cream BID; Test type: Superiority; response rate difference = -4.3, 95% CI 2-sided [-29.2 to 20.7], Standard Error of Mean 12.73 — The 95% confidence interval for the response rate difference was constructed from approximately normal distribution

2. Secondary Outcome: Change From Baseline in the Clinical Lichen Sclerosus Score (CLISSCO) at Week 12
Description: The CLISSCO is a validated tool to assess disease severity in vulvar lichen sclerosus. The Clinical Lichen Sclerosus Score consists of 12 items divided into 3 sections: symptoms (3 items; likely reversible [i.e., itch, pain, dysuria]); signs (3 items; possibly reversible [i.e., whitening, petechiae/ecchymosis, fissures]); and architectural changes (6 items; irreversible [i.e., skin fusion, perianal involvement, etc.]). All symptoms, signs, and architectural changes were rated on a 4-point Likert scale: 0 (absent), 1 (mild), 2 (moderate), and 3 (severe). The investigator documented the score of each of the 12 items; the CLISSCO was calculated by summing the score of each question, with a maximum score of 36 and a minimum score of 0. The higher the score, the more severe the disease. Additionally, the total score for each of the 3 sections (symptoms, signs, and architectural changes) was summarized by summing the scores of the questions in each section.
Time Frame: Baseline; Week 12
Population: ITT Population. Only participants with available data were analyzed. Mixed Model Repeated Measures (MMRM) model: response variable = treatment + visit + treatment by visit.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | DBVC Period: Ruxolitinib Cream 1.5% BID | DBVC Period: Vehicle Cream BID
Number analyzed (Participants) | 29 | 27
scores on a scale | -5.79 (0.80) | -3.03 (0.82)
Statistical Analysis 1: Comparison: DBVC Period: Ruxolitinib Cream 1.5% BID vs DBVC Period: Vehicle Cream BID; Test type: Superiority; p = 0.0188, Mixed Model Repeated Measures (MMRM); least squares mean difference = -2.76, 95% CI 2-sided [-5.05 to -0.47], Standard Error of Mean 1.14

3. Secondary Outcome: Change From Baseline in the Skin Pain NRS Score at Week 12
Description: Participants were instructed to complete and record the Skin Pain NRS in a diary each evening beginning on the day of screening through Week 12 or treatment discontinuation. Participants rated their pain, which included all types of pain (e.g., burning, tearing, pulling, stabbing, etc.) severity of lichen sclerosus by selecting a number from 0 (no pain) to 10 (worst imaginable pain) that best described the worst level of pain they experienced in the past 24 hours.
Time Frame: Baseline; Week 12
Population: ITT Population. Only participants with available data were analyzed. No imputation was performed for missing values. MMRM model: response variable = treatment + visit + treatment by visit.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | DBVC Period: Ruxolitinib Cream 1.5% BID | DBVC Period: Vehicle Cream BID
Number analyzed (Participants) | 29 | 26
scores on a scale | -3.22 (0.50) | -2.70 (0.52)
Statistical Analysis 1: Comparison: DBVC Period: Ruxolitinib Cream 1.5% BID vs DBVC Period: Vehicle Cream BID; Test type: Superiority; p = 0.4674, MMRM; least squares mean difference = -0.53, 95% CI 2-sided [-1.96 to 0.91], Standard Error of Mean 0.72

4. Secondary Outcome: Time to Achieve ITCH4
Description: as for outcome 1
Time Frame: up to 99.0 days
Population: ITT Population. Only those participants achieving a ≥4-point improvement in daily Itch NRS score from Baseline were analyzed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | DBVC Period: Ruxolitinib Cream 1.5% BID | DBVC Period: Vehicle Cream BID
Number analyzed (Participants) | 18 | 18
days | 35.0 [7.0 to 57.0] | 28.0 [6.0 to NA] — The upper limit of the confidence interval was not evaluable because there were too few participants with events.
Statistical Analysis 1: Comparison: DBVC Period: Ruxolitinib Cream 1.5% BID vs DBVC Period: Vehicle Cream BID; Test type: Superiority; p = 0.9072, Log Rank; Hazard Ratio (HR) = 0.970, 95% CI 2-sided [0.503 to 1.869] — Cox regression model was conducted to compare the difference in hazard rate

5. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE) During the Double-blind, Vehicle-controlled Period
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it is considered drug related. An AE could therefore have been any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study drug. A TEAE was defined as an AE either reported for the first time or the worsening of a pre-existing event after the first application of study drug.
Time Frame: from Baseline to Week 12 plus 30 days
Population: Safety Population: all participants who applied ruxolitinib 1.5% cream or vehicle cream at least once. Treatment groups for this population were determined according to the actual treatment the participant applied on Day 1 regardless of assigned treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | DBVC Period: Ruxolitinib Cream 1.5% BID | DBVC Period: Vehicle Cream BID
Number analyzed (Participants) | 31 | 30
Participants | 14 | 12

6. Secondary Outcome: Number of Participants With Any ≥Grade 3 TEAE During the Double-blind, Vehicle-controlled Period
Description: A TEAE was defined as an AE either reported for the first time or the worsening of a pre-existing event after the first application of study drug. The severity of AEs was assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 (v5.0) Grades 1 through 5. The investigator made an assessment of intensity for each AE and SAE reported during the study and assigned it to 1 of the following categories: Grade 1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; treatment not indicated. Grade 2: moderate; minimal, local, or noninvasive treatment indicated; limiting age-appropriate activities of daily living. Grade 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living. Grade 4: life-threatening consequences; urgent treatment indicated. Grade 5: fatal.
Time Frame: from Baseline to Week 12 plus 30 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DBVC Period: Ruxolitinib Cream 1.5% BID | DBVC Period: Vehicle Cream BID
Number analyzed (Participants) | 31 | 30
Participants | 1 | 0

7. Secondary Outcome: Number of Participants With Any TEAE During the Open-label Extension Period
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it is considered drug related. An AE could therefore have been any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study drug. A TEAE was defined as an AE either reported for the first time or the worsening of a pre-existing event after the first application of study drug.
Time Frame: from Week 12 to Week 24 plus 30 days
Population: Open-label Extension Evaluable Population: all participants who applied ruxolitinib 1.5% cream at least once during the Open-label Extension Period
Measure: Count of Participants; unit: Participants
Arm/Group | DBVC Period: Ruxolitinib Cream 1.5% BID | DBVC Period: Vehicle Cream BID
Number analyzed (Participants) | 29 | 27
Participants | 13 | 11

8. Secondary Outcome: Number of Participants With Any ≥Grade 3 TEAE During the Open-label Extension Period
Description: A TEAE was defined as an AE either reported for the first time or the worsening of a pre-existing event after the first application of study drug. The severity of AEs was assessed using the CTCAE v5.0 Grades 1 through 5. The investigator made an assessment of intensity for each AE and SAE reported during the study and assigned it to 1 of the following categories: Grade 1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; treatment not indicated. Grade 2: moderate; minimal, local, or noninvasive treatment indicated; limiting age-appropriate activities of daily living. Grade 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living. Grade 4: life-threatening consequences; urgent treatment indicated. Grade 5: fatal.
Time Frame: from Week 12 to Week 24 plus 30 days
Population: Open-label Extension Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | DBVC Period: Ruxolitinib Cream 1.5% BID | DBVC Period: Vehicle Cream BID
Number analyzed (Participants) | 29 | 27
Participants | 1 | 0

9. Secondary Outcome: Number of Participants With Any Clinically Meaningful Changes Over Time in Clinical Laboratory Test Results During the Double-blind, Vehicle-controlled Period
Description: The investigator determined if a clinical laboratory test value was clinically meaningful.
Time Frame: from Baseline to Week 12 plus 30 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DBVC Period: Ruxolitinib Cream 1.5% BID | DBVC Period: Vehicle Cream BID
Number analyzed (Participants) | 31 | 30
Participants | 0 | 0

10. Secondary Outcome: Number of Participants With Any Clinically Meaningful Changes Over Time in Vital Sign Values During the Double-blind, Vehicle-controlled Period
Description: The investigator determined if a clinical laboratory test value was clinically meaningful.
Time Frame: from Baseline to Week 12 plus 30 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DBVC Period: Ruxolitinib Cream 1.5% BID | DBVC Period: Vehicle Cream BID
Number analyzed (Participants) | 31 | 30
Participants | 0 | 0

11. Secondary Outcome: Number of Participants With Any Clinically Meaningful Changes Over Time in Clinical Laboratory Test Results During the Open-label Extension Period
Description: The investigator determined if a clinical laboratory test value was clinically meaningful.
Time Frame: from Week 12 to Week 24 plus 30 days
Population: Open-label Extension Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | DBVC Period: Ruxolitinib Cream 1.5% BID | DBVC Period: Vehicle Cream BID
Number analyzed (Participants) | 29 | 27
Participants | 0 | 0

12. Secondary Outcome: Number of Participants With Any Clinically Meaningful Changes Over Time in Vital Sign Values During the Open-label Extension Period
Description: The investigator determined if a clinical laboratory test value was clinically meaningful.
Time Frame: from Week 12 to Week 24 plus 30 days
Population: Open-label Extension Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | DBVC Period: Ruxolitinib Cream 1.5% BID | DBVC Period: Vehicle Cream BID
Number analyzed (Participants) | 29 | 27
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: up to approximately 32 weeks
Description: For safety analysis, participants who transitioned from treatment with vehicle to treatment with 1.5% BID ruxolitinib cream in the the Open-label Extension Period have been counted both in the vehicle arm and the ruxolitinib arm.
Groups:
- Ruxolitinib Cream 1.5% BID: Participants who completed the Week 12 assessments with no safety concerns, continued into the 12-week Open-label Extension Period, and applied ruxolitinib cream 1.5% BID for 12 weeks in the Open-label Extension Period.
- Vehicle Cream BID: Participants applied matching vehicle cream twice a day (BID) for 12 weeks in the Double-Blind Period.
Arm/Group | Ruxolitinib Cream 1.5% BID | Vehicle Cream BID
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/58 | 1/30
Other Adverse Events (participants affected / at risk) | 10/58 | 6/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ruxolitinib Cream 1.5% BID (N=58) | Vehicle Cream BID (N=30)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ruxolitinib Cream 1.5% BID (N=58) | Vehicle Cream BID (N=30)
COVID-19 (Infections and infestations) | 2 (2) | 2 (2)
Nasopharyngitis (Infections and infestations) | 3 (3) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 4 (5) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2023-12-18): https://cdn.clinicaltrials.gov/large-docs/45/NCT05593445/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-24): https://cdn.clinicaltrials.gov/large-docs/45/NCT05593445/SAP_001.pdf